CLINICAL TRIAL: NCT05446025
Title: MSH and CART Levels of Orexigenic Hormones (Which Increase Appetite), Orexin, Galanin and Anorexigenic Hormones (Which Reduce Appetite) in Patients With Hyperemesis Gravidarum
Brief Title: The Levels of the Orexin, Galanin and aMSH and CART in Patients With Hyperemesis Gravidarum
Status: Completed | Type: Observational
Sponsor: Siirt University (Other)
Responsible Party: Principal Investigator, Serif Aksin, Associate professor, Siirt University
Other Study IDs: SiirtUNIVers
Record Dates: First submitted 2022-06-26; First posted 2022-07-06 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Hyperemesis Gravidarum; Pregnancy Related
Keywords: vomiting; pregnant; ketonuria
MeSH Terms: conditions — Hyperemesis Gravidarum; Vomiting; Ketosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pregnant women with a diagnosis of hyperemesis gravidarum( n:50): Orexigenic hormones (appetizing) Orexin, galanin and anorexigenic hormones (decreasing appetite) aMSH and CART blood levels will be examined in patients with hyperemesis gravidarum.
  Interventions: Diagnostic Test: Blood sample
- Control group pregnants (n:50): Orexigenic hormones (appetizing) Orexin, galanin and anorexigenic hormones (decreasing appetite) aMSH and CART blood levels will be examined in the patients of the control group .
  Interventions: Diagnostic Test: Blood sample

INTERVENTIONS:
Diagnostic Test: Blood sample — Orexigenic hormones (appetizing) Orexin, galanin and anorexigenic hormones (decreasing appetite) aMSH and CART blood levels will be measured

SUMMARY:
Hyperemesis gravidarum is a disease of unknown etiology that is frequently encountered in pregnant women and seriously impairs their quality of life. In the United States, hyperemesis gravidarum is the most common cause of hospitalizations in the first half of pregnancy and is second only to preterm labor for hospitalizations during pregnancy overall. The prevalence of hyperemesis gravidarum is approximately 0.3-3% of pregnancies and varies due to different diagnostic criteria and ethnic differences in study populations. According to the latest guidelines from the American College of Obstetricians and Gynecologists (ACOG) on nausea and vomiting during pregnancy, there is still no single accepted definition for hyperemesis gravidarum. The most commonly cited criteria for the diagnosis of hyperemesis gravidarum include persistent, unrelated to other causes, ketonuria, electrolyte abnormalities and acid-base disturbances, as well as weight loss. Weight loss is usually stated as at least 5% loss. In normal individuals, the appetite regulation center is the hypothalamus. Neuropeptides released from hypothalamic neurons play an important role in the regulation of nutrition by acting both in the hypothalamus and other appetite-regulating centers in the brain. Among the neuropeptides that are secreted by the central nervous system and peripheral organs and also play an important role in the regulation of energy and appetite, there are neuropeptides known as orexigenic neuropeptides, which reduce energy expenditure and increase appetite, as well as anorexigenic neuropeptides, which, on the contrary, reduce appetite and increase energy expenditure. It is known that disorders in these pathways cause pathologies in appetite and food intake in normal individuals. In our study, we plan to examine the levels of some neuropeptides in patients with hyperemesis gravidarum in order to investigate whether these pathways are affected or not. In this study, we aimed to investigate whether orexigenic neuropeptides (Orexin, Galanin) and anorexigenic neuropeptides (aMSH, CART) levels are associated with hyperemesis gravidarum.

DETAILED DESCRIPTION:
Our aim in this study is to determine the levels of orexigenic and anorexigenic neuropeptides in patients with hyperemesis gravidarum and to determine whether there is a relationship between the function of the appetite center and the levels of these neuropeptides. For this purpose, approximately 50 pregnant women who were followed up with the diagnosis of hyperemesis gravidarum in Siirt Training and Research Hospital between 26 June 2022 and 30 october 2022 will be included in the study. The pregnant woman's age, pregnancy history, medical history will be recorded. Thyroid function test results, hemogram results and electrolyte levels of all patients will be recorded. Whole blood will be taken from these patients and the levels of Orexin and Galanin, which are orexigenic hormones, and aMSH and CART, which are anorexigenic hormones, will be checked. In the light of the information thus obtained, we plan to determine whether there is a relationship between hyperemesis gravidarum and the appetite center and between orexigenic and anorexigenic hormone levels.

ELIGIBILITY:
1-Inclusion Criteria:

5 to 20 weeks of pregnancy

Pregnants with a diagnosis of hyperemesis gravidarum

Pregnants who vomit more than 3 times a day

Those with 5 %more weight loss during pregnancy

detection of ketonuria

2-Exclusion Criteria:

food poisoning

Precision intestinal syndrome

Crohn's disease

Excessive alcohol consumption

Eating disorders such as anorexia and blomia

Neurological conditions such as meningitis, brain tumor and brain trauma

Migraine

Appendicitis

Chemotherapy drugs

Stomach and intestinal infections

Disorders such as celiac or lactose intolerance

-

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women diagnosed with hyperesis gravidarum
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-06-26 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Comparison of hyperemesis gravidarum and levels of orexigenic and anorexigenic blood hormones | Up to 20th week of gestation
  Orexigenic hormones (appetizing) Orexin, galanin and anorexigenic hormones (decreasing appetite) aMSH and CART blood levels will be examined in patients with hyperemesis gravidarum.(Blood hormones values will be measured by Elisa method(pg/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Şerif Aksin, Assoc.Prof, Study Director — Siirt University Medical Faculty Obstetrics and Gynecology Departmant
Locations (1):
- Siirt Üniversity Medical Faculty, Siirt, Turkey (Türkiye)

REFERENCES:
- [Background] Parker JA, Bloom SR. Hypothalamic neuropeptides and the regulation of appetite. Neuropharmacology. 2012 Jul;63(1):18-30. doi: 10.1016/j.neuropharm.2012.02.004. Epub 2012 Feb 19. PMID 22369786
- [Background] Sohn JW. Network of hypothalamic neurons that control appetite. BMB Rep. 2015 Apr;48(4):229-33. doi: 10.5483/bmbrep.2015.48.4.272. PMID 25560696
- [Background] London V, Grube S, Sherer DM, Abulafia O. Hyperemesis Gravidarum: A Review of Recent Literature. Pharmacology. 2017;100(3-4):161-171. doi: 10.1159/000477853. Epub 2017 Jun 23. PMID 28641304